CLINICAL TRIAL: NCT02354001
Title: Selective Estrogen Receptor Modulators (SERMs) - A Potential New Treatment for Women of Child-bearing Age With Psychotic Symptoms of Schizophrenia
Brief Title: Selective Estrogen Receptor Modulators for Women of Child-bearing Age With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Alfred (Other)
Collaborators: Monash University (Other)
Responsible Party: Principal Investigator, Jayashri Kulkarni, Professor, Professor, The Alfred
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 94/06
Record Dates: First submitted 2015-01-27; First posted 2015-02-03 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; mental illness; serm; raloxifene; clinical trial
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders | interventions — Raloxifene Hydrochloride; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Raloxifene Hydrochloride (Experimental): 120 mg per capsule (1 tablet daily)
  Interventions: Drug: Raloxifene hydrochloride
- placebo tablet (Placebo Comparator): 1 tablet daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Raloxifene hydrochloride — 120mg daily- 1 capsule for 12 week trial
  Other Names: Evista
  Arms: Raloxifene Hydrochloride
Drug: Placebo — 1 capsule daily for 12 week trial - lactose
  Other Names: Lactose
  Arms: placebo tablet

SUMMARY:
The aim of the project is to investigate the use of Raloxifene (a new form of estrogen) in the treatment of young women with schizophrenia and schizoaffective disorder. Raloxifene is a Selective Estrogen Receptor Modulator (SERM),which means that it can affect the central nervous system (CNS) effects of estrogen (eg. improving emotional symptoms, memory, information processing and concentration), without adversely affecting reproductive tissue/organs such as breast, uterus and ovaries. The investigators are conducting a double-blind, placebo controlled, three month study comparing the psychotic symptom response of women with schizophrenia in both groups. One group will receive standard antipsychotic medication plus 120mg Raloxifene, while the second group will receive standard antipsychotic medication plus oral placebo.

DETAILED DESCRIPTION:
Estrogen is hypothesised to be protective for women against early onset of severe symptoms of schizophrenia (Hafner, 1991; Seeman, 1992). This 'estrogen hypothesis' was derived from epidemiological, clinical and animal studies. Following the results of such studies, the investigators conducted a study (Kulkarni et al 1996) in which a group of premenopausal women with schizophrenia were given 0.02mg oral estradiol as an adjunct to antipsychotic drug treatment for eight weeks, and compared their progress with a similar group who received antipsychotic drugs only. The group receiving estrogen made a significantly more rapid recovery from acute psychotic symptoms and also reported improvement in their general health status. Subsequently, the investigators conducted a four week double-blind, placebo-controlled study, using 100mcg estradiol skin patches. The investigators found that the 12 premenopausal women who received the estradiol adjunct had a significantly lower total PANSS and BPRS score than 12 women who received placebo patches plus antipsychotic medication.

The major potential risks in using estrogen as a longer term adjunctive treatment in premenopausal women with schizophrenia appear to be the potential harmful effects of estrogen itself in its action on breast and uterine tissue.

Our studies were brief for this reason, in that the investigators used estrogen without progesterone over an eight week or four week period.

With the recent advent of Selective Estrogen Receptor Modulators, in particular Raloxifene Hydrochloride, there is the potential to harness the positive estrogenic effect on CNS neurotransmitter systems without affecting breast or uterine tissue. While the CNS effects of Raloxifene have not been fully studied, its actions are mediated through binding to estrogen receptors and can thereby regulate gene expression that is ligand, tissue or gene specific.

By inference then, Raloxifene would be expected to impact on dopamine and serotonin pathways in a similar fashion to conjugated estrogen. A study (Nickleisen et al 1999) on the effect of Raloxifene on cognition in healthy, postmenopausal women found a slight increase in verbal memory performance after one month of high dose treatment, while no other differences were found after 12 months of treatment. There are no studies in women with cognitive impairment where a treatment effect would be more likely to be apparent. Similarly, there are no clinical studies to date investigating the effect of Raloxifene on psychotic symptoms. To this end, the investigators are putting forward an investigator initiated clinical trial proposal to investigate the effect of adjunctive Raloxifene on psychotic symptoms in women with schizophrenia. This is, therefore, a study to follow our Pilot Study in the same area, but with an increase of Raloxifene from 60mg to 120mg daily.

ELIGIBILITY:
Inclusion Criteria:

* Physically well
* A current DSM-IV diagnosis of schizophrenia or related disorder.
* 18- 45 years
* Premenopausal (regular menstrual cycles and follicle stimulating hormone < 40 mIU/ml; for hysterectomised women, FSH< 40mIU/ml and estradiol> 120pmol/L)
* Able to give informed consent.
* PANSS total score > 60 (1 - 7 scale) and a score of 4 (moderate) or more on two or more of the following PANSS items: delusions, hallucinatory behaviour, conceptual disorganization or suspiciousness.
* No abnormality observed during physical breast examination.
* Documented normal PAP smear and pelvic examination in the preceding two years.

Exclusion Criteria:

* Patients with known abnormalities in the hypothalamo-pituitary gonadal axis, thyroid dysfunction, central nervous system tumours, active or past history of a venous thromboembolic event, or undiagnosed vaginal bleeding.
* Patients with any significant unstable medical illness such as epilepsy and diabetes or known active cardiac, renal or liver disease; presence of illness causing immobilisation.
* Patients whose psychotic illness is directly related to illicit substance use or who have a history of substance abuse or dependence during the last six months, or consumption of more than 30gm of alcohol (three standard drinks) per day.
* Smoking more than 20 cigarettes per day.
* Use of any form of estrogen, progestin or androgen as hormonal therapy, or antiandrogen including tibolone or use of phytoestrogen supplements as powder or tablet.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale (PANSS) | baseline and 12 weeks

SECONDARY OUTCOMES:
Change from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) score | baseline and 12 weeks
Change from baseline in Cognitive Test scores- MATRICS Consensus Cognitive Battery (MCCB) and Repeatable Battery for the Assessment of Neuropsychological Status Update (RBANS) | baseline and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Monash Alfred Psychiatry Research Centre, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Thomas N, Gurvich C, Hudaib AR, Gavrilidis E, Kulkarni J. Dissecting the syndrome of schizophrenia: Associations between symptomatology and hormone levels in women with schizophrenia. Psychiatry Res. 2019 Oct;280:112510. doi: 10.1016/j.psychres.2019.112510. Epub 2019 Aug 8. PMID 31415936